CLINICAL TRIAL: NCT03605238
Title: Clinical Study of CD19/CD20 tanCAR T Cells in Relapsed and/or Refractory AQP4-IgG Seropositive Neuromyelitis Optica Spectrum Disorders (NMOSD)
Brief Title: Treatment of Relapsed and/or Refractory AQP4-IgG Seropositive NMOSD by Tandem CAR T Cells Targeting CD19 and CD20
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: It was hard to recruit patients
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Wei Shihui, Professor of Neuro-Ophthalmology, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-NO-S2018-002-02
Record Dates: First submitted 2018-06-29; First posted 2018-07-30 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-08

CONDITIONS: Neuromyelitis Optica Spectrum Disorder
Keywords: Neuromyelitis Optica Spectrum Disorder; aquaporin4-IgG; CAR-T therapy
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Corticosteroids & tanCART19/20 (Experimental): Twelve days of high-dose IV methylprednisolone to reduce acute inflammation, then infuse anti-CD19/20-CAR retroviral vector-transduced autologous derived T cells only once.
  Interventions: Biological: Corticosteroids & tanCART19/20

INTERVENTIONS:
Biological: Corticosteroids & tanCART19/20 — Twelve days of high-dose IV methylprednisolone (1000mg×3 days, 500mg×3 days, 240mg×3 days, 120mg×3 days) before anti-CD19/20 CAR T cells infusion. The dose is 1E5~2E6 anti-CD19/20-CAR positive T cells. The cells infusion process may last for 30 min.

SUMMARY:
CAR-T therapy was proposed and has been recently used for cancer treatment. It has been hailed for its promising remission rates after early stage clinical trials for acute lymphoblastic leukemia. However, CAR-T therapy is seldom used for autoimmune diseases. Researchers only use it for the treatment of systemic lupus erythematosus (SLE). Neuromyelitis optica spectrum disorders (NMOSD), that include the neuromyelitis optica (NMO), are a group of inflammatory disorders of the central nervous system characterized by episodes of immune-mediated demyelination and axonal damage mainly involving optic nerves and spinal cord. NMO is characterized by the presence of an anti-Aquaporin-4 (AQP4) antibody, which can only be produced by differentiation of B cells to plasma cells. Because these anti-AQP4 antibodies may be pathogenic, B cells recognizing AQP4 may be directly involved in the disease process as well. B cells also play a role as potent antigen presenting cells in NMO. NMO has the characteristics of high recurrence rate and poor prognosis. In the conventional treatment options, NMOSD could be treated with corticosteroids and immunosuppressive drugs immunosuppressant (e.g. azathioprine, mycophenolate mofetil, rituximab). But these drugs could barely completely cure NMOSD. And now, chimeric antigen receptor modified T cell infusion maybe an effective treatment to solve these problems. The rationale for using CAR-T therapy in NMOSD is based on the known roles of B cells, antibody production and plasma cells in the pathophysiology of NMOSD. The strongest evidence of the importance of B cells in NMO comes from studies of B cell depletion, most commonly with anti-CD20 monoclonal antibody, rituximab. Emerging evidence indicates that peripheral B cells are activated during a relapse and plasmablast production of anti-AQP4 antibodies spikes. The investigators infuse tanCART19/20 to completely deplete B cells. The purpose of this study is to assess the safety and efficacy of this tanCART19/20 in the treatment of NMOSD.

DETAILED DESCRIPTION:
This study is being conducted to assess anti-CD19/20 CAR T cells safety and efficacy in treating patients with AQP4-IgG seropositive NMOSD.

PRIMARY OBJECTIVES:

I. To assess the safety of the tanCART-19/20 cells in treating NMOSD patients. II. Determine duration of in vivo survival of tanCART-19/20 cells.

SECONDARY OBJECTIVES:

I. To assess the efficacy of the tanCART-19/20 cells in treating NMOSD patients.

II. The secondary outcome measures: annual relapse rate (ARR), Expanded Disability Status Scale Score(EDDS), Best Corrected Visual Acuity (Log MAR), Spectral-Domain Optical Coherence Tomography (SD-OCT), Flash Visual Evoked Potential (FVEP) and Immunological assessments.

OUTLINE: Patients receive anti-CD19/20-CAR (coupled with CD137 and CD3 zeta signalling domains) vector-transduced autologous T cells on days 0 in the absence of unacceptable toxicity. The infusion dose is 1E5-2E6 CAR positive T cells/kg, and dose escalation methods obey the traditional 3+3 design (three doses groups: 1-2E5, 3-6E5, 1-2E6 CAR-T cells).

After completion of study treatment, patients are followed intensively for 6 months, every 6 months for 2 years, and annually thereafter for 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of neuromyelitis optica spectrum disorders (NMOSD) patients.
2. Patients with AQP4-IgG seropositive by cell-based assay.
3. Patients with corticosteroid treatment combined immunosuppressant (azathioprine or mycophenolate mofetil or rituximab) still recurrence.
4. Clinical evidence of at least 2 relapses in last 12 months or 3 relapses in the last 24 months with at least 1 relapse in the 12 months prior to the Screening.
5. Best corrected visual acuity(BCVA)<20/60.
6. Normal bone marrow reserve function: neutrophils>1 500/mm3, Hemoglobin > 10g/dL, Platelet count > 100 000/mm3.
7. Normal liver and kidney function: Creatinine < 2.5 mg/dl, ALT (alanine aminotransferase)/AST (aspartate aminotransferase) < 3x normal, Bilirubin < 2.0 mg/dl.
8. Successful test expansion of tanCART19/20 cells.
9. Adequate venous access for apheresis, and no other contraindications for leukapheresis.
10. Voluntary informed consent is given.

Exclusion Criteria:

1. Pregnant or lactating women (The safety of this therapy on unborn children is not known, Female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion).
2. Any serious, uncontrolled diseases (including, but not limit to, uncontrolled active infection, active hepatitis B or hepatitis C infection, HIV infection, unstable angina pectoris, congestive heart failure, serious arrhythmia).
3. Concurrent use of systemic steroids or immunosuppressant in the last two weeks.
4. Feasibility assessment during screening demonstrates < 30% transduction of target lymphocytes, or insufficient expansion (< 5-fold) in response to CD3/CD137 costimulation.
5. Other patients who are not suitable for CAR-T therapy judged by the biotherapy physician.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-15 (Estimated); Primary Completion 2019-08-15 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | From baseline to 12 months after
  defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events that are possibly, likely, or definitely related to study treatment.

SECONDARY OUTCOMES:
Annualized relapse rate (ARR) of NMOSD Attacks | Baseline, 12 months
  Compare annualized relapse rate before and one year after initial CAR-T administration.
Change in Expanded Disability Status Scale (EDDS) Score | Baseline, 12 months
  The EDSS is an ordinal clinical rating scale ranging from 0 (normal neurologic examination) to 10 (death) in half-point increments.
Change in Best Corrected Visual Acuity (Log MAR) | Baseline, 12 months
  Visual acuity assessment through Snellen's test chart.
Change in peripapillary retinal nerve fibre layer(pRNFL) | Baseline, 12 months
  Compared pRNFL before and one year after initial CAR-T administration.
Change in macular ganglion cell-inner plexiform layers (mGCIPL) | Baseline, 12 months
  Compared mGCIPL before and one year after initial CAR-T administration.
Change in Flash Visual Evoked Potential (FVEP) | Baseline, 12 months
  Compared FVEP before and one year after initial CAR-T administration.

OTHER OUTCOMES:
in vivo existence of tanCART19/20 | Baseline, 12 months
  RT-PCR (reverse transcription polymerase chain reaction) analysis of whole blood will be used to detect and quantify survival of tanCART-19/20 TCR (T-cell receptor) zeta:CD137 and TCR zeta cells over time.
Determination of serum immunoglobulins | Baseline, 12 months
  Compare serum IgG level before and one year after initial CAR-T administration.
Determination of serum AQP4 antibodies | Baseline, 12 months
  Compare serum AQP4-ab titers before and one year after initial CAR-T administration.
Determination of serum cytokines | Baseline, 12 months
  Compare serum cytokines before and one year after initial CAR-T administration.
Counts of peripheral blood B cell subsets | Baseline, 12 months
  Compare peripheral blood B cells before and one year after initial CAR-T administration.

CONTACTS AND LOCATIONS:
Overall Officials: Quangang Xu, PhD, Study Director — Chinese PLA General Hospital; Huanfen Zhou, PhD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- People's Liberation of Army General Hospital (PLAGH), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No